CLINICAL TRIAL: NCT01797159
Title: "A Phase II Trial of Hippocampal-Sparing Cranial Irradiation (PCI) for Small-Cell Lung Cancer (SCLC)"
Brief Title: Hippocampal Prophylactic Cranial Irradiation for Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J12127; NA_00078659 (Other: JHMIRB)
Record Dates: First submitted 2012-11-30; First posted 2013-02-22 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Small-cell Lung Cancer; SCLC; Small Cell Lung Cancer Limited Stage
Keywords: Prophylactic Cranial Irradiation; PCI; Hippocampal-sparing irradiation
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hippocampal-sparing PCI (Experimental): Hippocampal-sparing PCI 25 Gy in 10 fractions
  Interventions: Radiation: Hippocampal-sparing Prophylactic Cranial Irradiation

INTERVENTIONS:
Radiation: Hippocampal-sparing Prophylactic Cranial Irradiation — Hippocampal-sparing Prophylactic Cranial Irradiation

SUMMARY:
The Investigators are looking to compare standard treatment for the management of small cell lung cancer (SCLC) which is prophylactic cranial Irradiation (PCI) (shown to be very good in patient survival) with cranial sparing PCI. Although standard of care PCI is successful in patient survival it also has neurologic side-effects. The Investigators are hoping the cranial sparing PCI has the same positive survival results with the added benefit of lowering neurological side-effects.

DETAILED DESCRIPTION:
The standard of care in management of small cell lung cancer consists of chemotherapy plus thoracic radiation followed by prophylactic cranial irradiation (PCI) based on a randomized trial that demonstrated a significant improvement in overall survival (OS) with PCI. Unfortunately radiation therapy to the brain is associated with neurocognitive toxicity, which may be at least in part related to radiation induced injury to neural progenitor cells in the hippocampus. Both human and animal data suggest an inverse relationship between radiation dose to the hippocampus and performance on neuropsychological testing. We hypothesize that hippocampal sparing PCI will allow improved performance on tests of short term memory and executive function compared to a historical control (RTOG 0212) receiving the same dose of conventional PCI. The primary objective of this study is to evaluate performance on the Hopkins Verbal Learning Test-Revised for delayed recall at 6 months following hippocampal-sparing PCI relative to the historical control. Secondary objectives are to estimate: 1) composite cognitive function following hippocampal-sparing PCI relative to the historical control and 2) the rate of metastases in the hippocampus at 2 years following hippocampal-sparing PCI. The long term goal of this research is to reduce the long term sequelae of radiation therapy for both primary and metastatic brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have newly diagnosed and confirmed small-cell lung cancer (SCLC)
* Patient must have a performance status of 1 or higher
* Patients must not have received previous irradiation to the brain
* Patients must have limited stage disease with complete response to chemotherapy and consolidative chest radiotherapy that was documented at least on standard chest x-rays within one month of study entry
* Negative MRI or CT scan of the brain at least one month before protocol entry
* Women of child-bearing potential must have a negative pregnancy test and also agree to use adequate contraceptives while on protocol
* Patient must be able to understand and sign the informed consent document
* Patient must be informed of the investigational aspect to this trial prior to singing the informed consent document

Exclusion Criteria:

* Patients receiving prior external beam irradiation to the head or neck, including any form of stereotactic irradiation
* Radiographic evidence of brain metastases and/or ipsilateral lung metastases/malignant pleural effusion
* Planned concurrent chemotherapy or antitumoral agent during PCI
* Concomitant malignancy or malignancy within the past five years other than nonmelanomatous skin cancer or carcinoma in situ of the cervix
* Patients with minimal pleural effusion evident on chest X-ray; minimal pleural effusion visible on chest CT is allowed.
* Patients with epilepsy requiring permanent oral medication
* Patients must not have a serious medical or psychiatric illness that would, in the opinion of the investigator, prevent informed consent or completion of protocol treatment, and/or follow-up visits.
* Patients may not take Memantine. This is the only eligibility criterion that has been added to those of RTOG 0212, since some physicians might now prescribe Memantine. This medication would not have been given at the time of enrollment on RTOG 0212 and its administration could confound the results of this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03-11 (Actual); Primary Completion 2018-03-18 (Actual); Study Completion 2019-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Redmond, M.D., Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Bayview Medical Center, Baltimore, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data with PIs who are not included on the study team.

REFERENCES:
- [Derived] Redmond KJ, Hales RK, Anderson-Keightly H, Zhou XC, Kummerlowe M, Sair HI, Duhon M, Kleinberg L, Rosner GL, Vannorsdall T. Prospective Study of Hippocampal-Sparing Prophylactic Cranial Irradiation in Limited-Stage Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2017 Jul 1;98(3):603-611. doi: 10.1016/j.ijrobp.2017.03.009. Epub 2017 Mar 14. PMID 28581401

RESULTS

PARTICIPANT FLOW:
Groups:
- Hippocampal-sparing PCI: Hippocampal-sparing Prophylactic Cranial Irradiation (PCI) 25 Gy in 10 fractions
Period: Overall Study
Arm/Group | Hippocampal-sparing PCI
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Hippocampal-sparing PCI: Hippocampal-sparing PCI 25 Gy in 10 fractions
  Hippocampal-sparing Prophylactic Cranial Irradiation
Arm/Group | Hippocampal-sparing PCI
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 61 [38 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Effect of Hippocampal-sparing Prophylactic Cranial Irradiation (PCI) on Possible Delayed Recall Toxicity as Assessed by the Hopkins Verbal Learning Test-Revised (HVLT-R) for Delayed Recall
Description: The primary endpoint of this study is cognitive function or memory. Memory is measured by participant performance on the Hopkins Verbal Learning Test-Revised for delayed recall (HVLT-R-Delayed Recall) at 6 months following hippocampal-sparing PCI. The HVLT-Delayed minimum and Maximum scores are 0-12. A higher score means a better outcome.
Time Frame: Baseline, 6 months and 12 months post radiation treatment
Population: At the 6 month timepoint, only 17 participants completed the test, and at the 12 month time point only 14 participants took the test.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hippocampal-sparing PCI
Number analyzed (Participants) | 20
score on a scale
  Baseline | 7.45 (2.64)
  6 months: number analyzed (Participants) | 17
  6 months | 7.06 (2.77)
  12 months: number analyzed (Participants) | 14
  12 months | 7.36 (2.87)

2. Secondary Outcome: Compare Cognitive Function Following Sparing PCI to That of Standard PCI
Description: Composite cognitive function following hippocampal-sparing PCI relative to a historical control receiving standard PCI.
  HVLT-R Hopkins Verbal Learning Test Revised and Brief Visuospatial Memory Test-Revised (BVMT-R)
  * Total Recall (0-36) higher = better
  * Delayed Recall (0-12) higher = better
  * Discrimination (-12 to 12) higher = better Trail Making A & B (0-300 seconds) higher = poorer Controlled Oral Word Association (COWA) (0-180) higher = better Mini-Mental State Exam (MMSE) (0-30) higher = better Perceptual Comparison Test (PCT) (0-128) higher = better Brief Test of Attention (BTA) (0-20) higher = better Calibrated Ideational Fluency Assessment (CIFA)
  * Letter Word Fluency (0-120) higher = better
  * Category Word Fluency (0-120) higher = better
  * Verbal Fluency (0-240) higher = better Learning and Memory
  * Verbal Composite T score (mean = 100, standard deviation = 15), higher = better
  * Visual Composite T score (mean = 100, standard deviation = 15), higher = better
Time Frame: Baseline
Population: Data is presented for Hippocampal-sparing PCI (from this study). 19 participants completed the test at baseline. No data from standard PCI for comparison to be done.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hippocampal-sparing PCI
Number analyzed (Participants) | 19
score on a scale
  HVLT-R Total Recall | 23.2 (3.35)
  HVLT-R Delayed Recall | 7.45 (2.64)
  HVLT-R Discrimination | 10.75 (1.25)
  Trail Making A | 30.1 (9.79)
  Trail Making B | 89.7 (59)
  COWA | 32.4 (13.7)
  MMSE | 28.3 (1.05)
  PCT | 59.1 (13.7)
  BTA | 16.2 (2.93)
  CIFA: Letter Word Fluency | 25.3 (7.75)
  CIFA: Category Word Fluency | 44.2 (8.39)
  CIFA: Verbal Fluency | 68.9 (12.3)
  BVMT-R Total Recall | 19.7 (7.9)
  BVMT-R Delayed Recall | 8.63 (4.62)
  BVMT-R Discrimination | 5.74 (.562)
  Learning and Memory: Verbal | 93.2 (15.2)
  Learning and Memory: Visual | 96.4 (23.7)

3. Secondary Outcome: Compare Cognitive Function Following Sparing PCI to That of Standard PCI
Description: as for outcome 2
Time Frame: 6 months post radiation treatment
Population: Data is presented for Hippocampal-sparing PCI (from this study). 14 participants completed the test at 6 months. No data from standard PCI for comparison to be done.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hippocampal-sparing PCI
Number analyzed (Participants) | 14
score on a scale
  HVLT-R Total Recall | 23.6 (5.44)
  HVLT-R Delayed Recall | 7.06 (2.77)
  HVLT-R Discrimination | 11.1 (4.76)
  Trail Making A | 34.0 (10.3)
  Trail Making B | 101 (69.5)
  COWA | 31.4 (13.1)
  MMSE | 27.2 (2.10)
  PCT | 54.9 (15)
  BTA | 15.1 (3.22)
  CIFA: Letter Word Fluency | 24.1 (10.7)
  CIFA: Category Word Fluency | 40.9 (10.1)
  CIFA: Verbal Fluency | 65.1 (19.9)
  BVMT-R Total Recall | 18.7 (6.5)
  BVMT-R Delayed Recall | 7.64 (2.28)
  BVMT-R Discrimination | 5.64 (1.08)
  Learning and Memory: Verbal | 95.4 (18)
  Learning and Memory: Visual | 96.0 (16.1)

4. Secondary Outcome: Compare Cognitive Function Following Sparing PCI to That of Standard PCI
Description: as for outcome 2
Time Frame: 12 months post radiation treatment
Population: Data is presented for Hippocampal-sparing PCI (from this study). 14 participants completed the test at 12 months. No data from standard PCI for comparison to be done.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hippocampal-sparing PCI
Number analyzed (Participants) | 14
score on a scale
  HVLT-R Total Recall | 21.5 (4.94)
  HVLT-R Delayed Recall | 7.36 (2.87)
  HVLT-R Discrimination | 10.6 (1.22)
  Trail Making A | 29.6 (10.3)
  Trail Making B | 101.2 (72.3)
  COWA | 34.2 (13.5)
  MMSE | 27.7 (1.7)
  PCT | 55.6 (18.8)
  BTA | 14.7 (4.31)
  CIFA: Letter Word Fluency | 25.1 (8.88)
  CIFA: Category Word Fluency | 42.5 (7.78)
  CIFA: Verbal Fluency | 66.9 (14.1)
  BVMT-R Total Recall | 19.1 (6.29)
  BVMT-R Delayed Recall | 7.50 (2.38)
  BVMT-R Discrimination | 5.71 (0.611)
  Learning and Memory: Verbal | 92.8 (17.7)
  Learning and Memory: Visual | 94.4 (17.5)

5. Secondary Outcome: Compare Change in Quality of Life of Hippocampal-sparing PCI Treatment Outcome to Standard PCI Treatment Quality of Life Questionnaire (QLQ)-C30
Description: Evaluate quality of life following hippocampal-sparing PCI relative to historical control receiving standard PCI. Difference between 6 months and baseline.
  Questions on the Quality of Life Questionnaire (QLQ-C30) assessment are on a four-point scale from "not at all" to "very much". Raw scores are linearly converted to a 0-100 scale with higher scores reflecting higher levels of function and higher levels of symptom burden. Questions on the QLQ-C30 cover the following:
  * Dyspnoea
  * Insomnia
  * Appetite
  * Constipation
  * Diarrhoea
  * Finances
  * Fatigue
  * Nausea/Vomiting
  * Pain
  * Physical Function
  * Role Function
  * Emotional Function
  * Cognitive Function
  * Social Function
  * Global QoL
Time Frame: Baseline and 6 months post radiation treatment
Population: Data is presented for Hippocampal-sparing PCI (from this study). No data from standard PCI for comparison to be done.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hippocampal-sparing PCI
Number analyzed (Participants) | 20
score on a scale
  Dyspnoea | 11.1 (30)
  Insomnia | -9.5 (30.5)
  Appetite | 20 (32.9)
  Constipation | 6.7 (44)
  Diarrhoea | 0 (12.6)
  Finances | 2.4 (35.7)
  Fatigue | 14.1 (26.4)
  Nausea/Vomiting | 3.3 (25.4)
  Pain | 2.2 (31.4)
  Physical Function | -11.6 (19.8)
  Role Function | -4.4 (23.1)
  Emotional Function | 0 (22)
  Cognitive Function | 11.1 (16.3)
  Social Function | 8.9 (35)
  Global QoL | -5.2 (26.3)

6. Secondary Outcome: Compare Change in Quality of Life of Hippocampal-sparing PCI Treatment Outcome to Standard PCI Treatment QLQ-C30
Description: Evaluate quality of life following hippocampal-sparing PCI relative to historical control receiving standard PCI. Difference between 12 months and baseline.
  Questions on the Quality of Life Questionnaire (QLQ-C30) assessment are on a four-point scale from "not at all" to "very much". Raw scores are linearly converted to a 0-100 scale with higher scores reflecting higher levels of function and higher levels of symptom burden. Questions on the QLQ-C30 cover the following:
  * Dyspnoea
  * Insomnia
  * Appetite
  * Constipation
  * Diarrhoea
  * Finances
  * Fatigue
  * Nausea/Vomiting
  * Pain
  * Physical Function
  * Role Function
  * Emotional Function
  * Cognitive Function
  * Social Function
  * Global QoL
Time Frame: Baseline and 12 months post radiation treatment
Population: Data is presented for Hippocampal-sparing PCI (from this study). No data from standard PCI for comparison to be done.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hippocampal-sparing PCI
Number analyzed (Participants) | 20
score on a scale
  Dyspnoea | 2.8 (26.4)
  Insomnia | -5.6 (31.2)
  Appetite | -3 (10)
  Constipation | 0 (47.1)
  Diarrhoea | 2.8 (17.2)
  Finances | 2.8 (22.3)
  Fatigue | -0.9 (21.9)
  Nausea/Vomiting | -1.4 (26.1)
  Pain | 2.8 (19.9)
  Physical Function | -4.8 (17.9)
  Role Function | 0 (22.5)
  Emotional Function | 5.6 (14.8)
  Cognitive Function | -9.7 (20.7)
  Social Function | 9.7 (23)
  Global QoL | 2.1 (15.9)

7. Secondary Outcome: Compare Change in Quality of Life of Hippocampal-sparing PCI Treatment Outcome to Standard PCI Treatment Quality of Life Questionnaire-Brain Cancer (QLQ-BN20)
Description: Evaluate quality of life following hippocampal-sparing PCI relative to historical control receiving standard PCI. Difference between 6 months and baseline.
  Questions on the Quality of Life Questionnaire-Brain Cancer (QLQ-BN20) are rated on a four-point scale ('not at all', 'a little', 'quite a bit' and 'very much'), and are linearly transformed to a 0-100 scale. Higher scores represent more severe symptoms. Questions on the QLQ-BN20 cover the following:
  * Headaches
  * Seizures
  * Drowsy
  * Hair loss
  * Itching
  * Weakness
  * Bladder
  * Future Uncertainty
  * Visual Disorder
  * Motor Dysfunction
  * Communication Deficit
Time Frame: Baseline and 6 months post radiation treatment
Population: Data is presented for Hippocampal-sparing PCI (from this study). No data from standard PCI for comparison to be done.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hippocampal-sparing PCI
Number analyzed (Participants) | 20
score on a scale
  Headaches | 13.3 (32.9)
  Seizures | -4.4 (17.2)
  Drowsy | 0 (25.2)
  Hair loss | 2.2 (29.5)
  Itching | 6.7 (28.7)
  Weakness | 13.3 (24.6)
  Bladder | 11.1 (20.6)
  Future Uncertainty | 0.6 (27)
  Visual Disorder | 6.3 (17.3)
  Motor Dysfunction | 7.1 (22.5)
  Communication Deficit | 12.7 (10.5)

8. Secondary Outcome: Compare Change in Quality of Life of Hippocampal-sparing PCI Treatment Outcome to Standard PCI Treatment Using the Quality of Life Questionnaire-Brain Cancer (QLQ-BN20).
Description: Evaluate quality of life following hippocampal-sparing PCI relative to historical control receiving standard PCI. Difference between 12 months and baseline.
  Questions on the Quality of Life Questionnaire-Brain Cancer (QLQ-BN20) are rated on a four-point scale ('not at all', 'a little', 'quite a bit' and 'very much'), and are linearly transformed to a 0-100 scale. Higher scores represent more severe symptoms. Questions on the QLQ-BN20 cover the following:
  * Headaches
  * Seizures
  * Drowsy
  * Hair loss
  * Itching
  * Weakness
  * Bladder
  * Future Uncertainty
  * Visual Disorder
  * Motor Dysfunction
  * Communication Deficit
  Headaches Seizures Drowsy Hair loss Itching Weakness Bladder Future Uncertainty Scale Visual Disorder Scale Motor Dysfunction Scale Communication Deficit Scale
Time Frame: Baseline and 12 months post radiation treatment
Population: Data is presented for Hippocampal-sparing PCI (from this study). No data from standard PCI for comparison to be done.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hippocampal-sparing PCI
Number analyzed (Participants) | 20
score on a scale
  Headaches | 9.1 (33.6)
  Seizures | -3 (10.1)
  Drowsy | -6.1 (29.1)
  Hair loss | -15.2 (22.9)
  Itching | 9.1 (15.6)
  Weakness | 6.1 (29.1)
  Bladder | 12.1 (30.8)
  Future Uncertainty | -3 (23.9)
  Visual Disorder | 3 (17.3)
  Motor Dysfunction | 6.7 (17.5)
  Communication Deficit | 6.7 (11.9)

9. Secondary Outcome: Number Participants With Hippocampus Brain Metastases Following Sparing PCI
Description: The number of participants with brain metastases after sparing PCI treatment was assessed to be compared to two existing studies.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hippocampal-sparing PCI
Number analyzed (Participants) | 20
Participants | 4

10. Secondary Outcome: Assess if Development of Leptomeningeal Carcinomatosis Following Sparing PCI is Higher Than Expected
Description: Determine whether development of leptomeningeal carcinomatosis following hippocampal-sparing PCI is higher than expected.
Time Frame: 6 months, 12 months, 18 months and 24 months post radiation treatment
Population: Data for this outcome measure was not collected.
Arm/Group | Hippocampal-sparing PCI
Number analyzed (Participants) | 0

11. Secondary Outcome: Percentage of Participants Surviving Following Hippocampal-sparing PCI
Description: To evaluate the survival rates of study participants following hippocampal-sparing PCI.
Time Frame: Up to 24 months post radiation treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hippocampal-sparing PCI
Number analyzed (Participants) | 20
percentage of participants | 88 [68 to 100]

ADVERSE EVENTS:
Time Frame: Adverse events were followed for a one-year period.
Arm/Group | Hippocampal-sparing PCI
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hippocampal-sparing PCI (N=20)
Fatigue (General disorders) | 18
Alopecia (General disorders) | 14
cough (Respiratory, thoracic and mediastinal disorders) | 15
Dsypnea (Respiratory, thoracic and mediastinal disorders) | 11
Dysphagia (General disorders) | 9
Anorexia (General disorders) | 7
Nausea (Gastrointestinal disorders) | 7
Tinnitus (Ear and labyrinth disorders) | 7
Memory Loss (General disorders) | 7
Insomnia (General disorders) | 11
Taste Disturbance (General disorders) | 6
Pain due to radiation therapy (Surgical and medical procedures) | 6
Constipation (Gastrointestinal disorders) | 6
Skin (Skin and subcutaneous tissue disorders) | 6
Mucus (General disorders) | 6
Dermatitis (Skin and subcutaneous tissue disorders) | 6
Dizziness/lightheaded (General disorders) | 5
Vomit (Gastrointestinal disorders) | 5
Pharynx and esophogus (Respiratory, thoracic and mediastinal disorders) | 4
Dysgeusia (General disorders) | 3
Headache (General disorders) | 3
Neuropathy (Nervous system disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 11
Ocular Visual (Eye disorders) | 3
Personality Behavioral (Psychiatric disorders) | 4
Hearing Changes (Ear and labyrinth disorders) | 3
Hot Flash (General disorders) | 2
Urinary Incontinence (Renal and urinary disorders) | 2
Voice changes (General disorders) | 2
Aphasia (Nervous system disorders) | 2
Pain (General disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT01797159/Prot_SAP_000.pdf